CLINICAL TRIAL: NCT02279719
Title: A Phase Ib/II Clinical Study of BBI608 in Combination With Sorafenib, or BBI503 in Combination With Sorafenib in Adult Patients With Hepatocellular Carcinoma
Brief Title: A Study of BBI608 in Combination With Sorafenib, or BBI503 in Combination With Sorafenib in Adult Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBIHCC-103; BBI608-503-103HCC (Other: Boston Biomedical, Inc.)
Record Dates: First submitted 2014-10-24; First posted 2014-10-31 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — napabucasin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BBI608 and Sorafenib (Experimental)
  Interventions: Drug: BBI608; Drug: Sorafenib
- BBI503 and Sorafenib (Experimental)
  Interventions: Drug: BBI503; Drug: Sorafenib
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: BBI608 — BBI608 will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study.
  Other Names: Napabucasin; BBI-608; BB608
  Arms: BBI608 and Sorafenib
Drug: BBI503 — BBI503 will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study.
  Other Names: Amcasertib; BBI-503; BB503
  Arms: BBI503 and Sorafenib
Drug: Sorafenib — Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
  Other Names: Nexavar

SUMMARY:
This is an open label, three-arm, phase 1 dose escalation study and phase 2 study of BBI608 in combination with sorafenib, or BBI503 in combination with sorafenib. The study population is adult patients with advanced hepatocellular carcinoma who have not received systemic chemotherapy.

DETAILED DESCRIPTION:
This is an open label, three-arm, phase 1 dose escalation study and phase 2 study of BBI608 in combination with sorafenib, or BBI503 in combination with sorafenib. The study population is adult patients with advanced hepatocellular carcinoma (HCC) who have not received systemic chemotherapy.

The phase 1 portion will involve dose-escalation of BBI608 administered in combination with a fixed starting dose of sorafenib (Arm 1), and dose escalation of BBI503 administered in combination with a fixed starting dose of sorafenib (Arm 2). The fixed starting dose-level of sorafenib for both arms will be 400 mg twice daily (800 mg total daily dose). Eligible patients will be randomized to either Arm 1 or Arm 2.

The phase 2 portion will be an open-label, 3-arm, randomized trial of patients with advanced HCC who have not received prior systemic treatment. Patients will be randomized to receive either, Arm 1: sorafenib administered in combination with BBI608 (at the RP2D determined for BBI608 plus sorafenib during the phase 1 portion); Arm 2: sorafenib in combination with BBI503 (at the RP2D determined for BBI503 plus sorafenib during the phase 1 portion), or Arm 3: sorafenib alone at a starting dose of 400 mg twice daily. The starting dose for sorafenib is the same for all study arms.

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH) and local regulatory requirements
2. Histologically or cytologically confirmed hepatocellular carcinoma that is metastatic, unresectable, or recurrent.

   1. Patients must not be candidates for curative resection
   2. Patients who have recurrent disease after having had one or more prior resections may be eligible, provided that they are not candidates for further curative resection.
   3. Patients who have recurrent hepatocellular carcinoma following hepatic transplantation are excluded unless the following criteria are met:

   i. Transplantation was performed at least 6 months prior to the relapse of HCC. ii. Patients are on stable immune suppressive therapy with no clinical evidence of rejection.

   iii. Are receiving ≤ 2.5 mg everolimus daily. d. Patients with known HIV infection are excluded. e. Patients with Hepatitis B are eligible provided there is no active viral replication. Patients with Hepatitis C who are not on interferon are eligible.
3. Patients who have a diagnosis of hepatocellular carcinoma made through radiologic imaging may be eligible, provided they meet the criteria according to the American Association for the Study of Liver Disease, AASLD (Bruix and Sherman, 2005; Bruix and Sherman, 2011)
4. Patients must be candidates for sorafenib
5. Must have had no previous systemic anti-cancer treatment, though previous loco-regional therapy is allowed:

   a. Prior treatment with any of the following is allowed: trans-arterial embolization, trans-arterial chemo-embolization, percutaneous ethanol injection, radio-embolization, radio-frequency ablation, or other ablation techniques.
6. Must be Child-Pugh class A

   a. Patients with uncontrolled massive ascites or presence of hepatic encephalopathy are excluded
7. Must have total serum bilirubin ≤ 3 mg/dl
8. ≥ 18 years of age
9. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
11. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 or BBI503 dose
12. Females of childbearing potential must have a negative serum pregnancy test
13. Aspartate Aminotransferase (AST) and Alanine transaminase (ALT) < 5.0x the upper limit of normal (ULN)
14. Glomerular filtration rate (GFR) > 45 mL/min/1.73m^2 according to the Cockcroft-Gault estimation.

13. Hemoglobin ≥ 8.5 mg/dl 14. Absolute neutrophil count ≥ 1.5 x 10^9/L 15. Platelets ≥ 75 x 10^9/L 16. Life expectancy ≥ 3 months

Exclusion Criteria

1. Previous treatment with sorafenib
2. Patients with known hypersensitivity to sorafenib or any other component of sorafenib.
3. Previous systemic anti-vascular endothelial growth factor (VEGF) or any prior systemic anti-cancer therapy, including prior treatment with systemic agents such as regorafenib, ramucirumab, pazopanib, or experimental agents such as brivanib.
4. Have had a surgical procedure requiring general anesthesia or inpatient hospitalization for recovery less than 4 weeks prior to beginning protocol therapy.
5. Have had a loco-regional procedure for the treatment of hepatocellular carcinoma (such as a percutaneous, trans-arterial, or radio-ablative procedure) less than 4 weeks prior to beginning protocol therapy. Protocol therapy may begin a minimum of 4 weeks after such a procedure provided the following criteria are met:

   1. There is progression of disease documented by RECIST 1.1
   2. All adverse events from the procedure have resolved or have been deemed irreversible and the patient meets inclusion criteria.
6. Any known symptomatic or untreated brain metastases requiring increase of steroid dose within 2 weeks prior to starting on study. Patients with treated brain metastases must be stable for 4 weeks after completion of that treatment. Patients must have no clinical symptoms from brain metastases and must be either off steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated.
7. Pregnant or breastfeeding
8. Significant gastrointestinal disorder(s), (e.g., Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection) such that, in the opinion of the treating investigator, absorption of oral medications may be impaired.
9. Unable or unwilling to swallow BBI608, BBI503, or sorafenib capsules or tablets
10. Uncontrolled inter-current illness including, but not limited to: ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), or uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements (e.g. no reliable transportation).
11. Subjects with a history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present that, in the opinion of the investigator, will not affect patient outcome in the setting of current hepatocellular carcinoma diagnosis.
12. Abnormal ECGs which are clinically significant such as QT prolongation (QTc > 480 msec), clinically significant cardiac enlargement or hypertrophy, new bundle branch block, or signs of active ischemia. Patients with evidence of prior infarction who are New York Heart Association (NYHA) functional classes II, III, or IV are excluded, as are patients with marked arrhythmias such as Wolff Parkinson White pattern or complete atrioventricular (AV) dissociation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-12; Primary Completion 2019-07 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Southern California Research Center, Coronado, California
  - California Center Associates for Research and Excellence, Inc. (Ccare), Encinitas, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USOR - Rocky Mountain Cancer Centers, Denver, Colorado
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Piedmont Cancer Institute, P.C., Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Kansas City Research Institure, Kansas City, Missouri
  - USOR - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - The Valley Hospital Luckow Pavilion, Paramus, New Jersey
  - USOR - New York Oncology Hematology, Albany, New York
  - University of Rochester, Wilmot Cancer Institute, Rochester, New York
  - Carolinas Health Care System, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Vontz Center, Cincinnati, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - USOR - Texas Oncology, Austin Midtown, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Joe Battle, El Paso, Texas
  - USOR - Texas Oncology, Fort Worth 12th Ave, Fort Worth, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology-McAllen South Second Street, McAllen, Texas
  - USOR - Texas Oncology, Tyler, Tyler, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Napabucasin+Sorafenib Phase IB Dose- Level 1: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin will be 160 mg twice daily Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Napabucasin+Sorafenib Phase IB Dose-Level 2: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin will be 240 mg twice daily Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasertib +Sorafenib Phase IB Dose- Level 1: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 100mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasertib+Sorafenib Phase IB Dose-Level 2: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 200mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Napabucasin+Sorafenib Phase II: Phase II Napabucasin will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasertib+Sorafenib Phase II: Phase II Amcasertib will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Sorafenib Phase II: Phase II Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
Period: Overall Study
Arm/Group | Experimental Napabucasin+Sorafenib Phase IB Dose- Level 1 | Experimental Napabucasin+Sorafenib Phase IB Dose-Level 2 | Experimental Amcasertib +Sorafenib Phase IB Dose- Level 1 | Experimental Amcasertib+Sorafenib Phase IB Dose-Level 2 | Experimental Napabucasin+Sorafenib Phase II | Experimental Amcasertib+Sorafenib Phase II | Sorafenib Phase II
Started | 5 | 10 | 4 | 9 | 28 | 10 | 31
Completed | 5 | 10 | 4 | 9 | 25 | 10 | 28
Not Completed | 0 | 0 | 0 | 0 | 3 | 0 | 3
Not completed — Patients randomized but never treated | 0 | 0 | 0 | 0 | 3 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Experimental Napabucasin +Sorafenib Phase IB- Dose Level 1: Napabucasin will be administered orally twice daily in combination with sorafenib.
  The dose of Napabucasin will be 160 mg twice daily Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Napabucasin +Sorafenib Phase IB- Dose Level 2: Napabucasin will be administered orally twice daily in combination with sorafenib.
  The dose of Napabucasin will be 240 mg twice daily Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasertib +Sorafenib Phase IB- Dose Level 1: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 100mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug
- Experimental Amcasertib +Sorafenib Phase IB- Dose Level 2: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 200mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Napabucasin +Sorafenib Phase II: Phase II Napabucasin will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasertib +Sorafenib Phase II: Phase II Amcasertib will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Experimental Napabucasin +Sorafenib Phase IB- Dose Level 1 | Experimental Napabucasin +Sorafenib Phase IB- Dose Level 2 | Experimental Amcasertib +Sorafenib Phase IB- Dose Level 1 | Experimental Amcasertib +Sorafenib Phase IB- Dose Level 2 | Experimental Napabucasin +Sorafenib Phase II | Experimental Amcasertib +Sorafenib Phase II | Sorafenib Phase II | Total
Number analyzed (Participants) | 5 | 10 | 4 | 9 | 28 | 10 | 31 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (5.22) | 70.8 (4.42) | 55.0 (22.20) | 60.6 (5.22) | 64.1 (8.72) | 68.4 (9.98) | 67.7 (8.73) | 65.7 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 3 | 4 | 3 | 7 | 21
  Male | 4 | 9 | 2 | 6 | 24 | 7 | 24 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 1 | 2 | 0 | 9 | 13
  White | 5 | 9 | 2 | 5 | 18 | 8 | 19 | 66
  More than one race | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Dose Limiting Toxicities for the Napabucasin and Amcasertib Arm in Combination With Sorafenib for Phase IB
Description: To assess the dose limiting toxicities for phase IB
Time Frame: 16 weeks including 2-week Sorafenib run-in period prior to initiation of combination therapy
Measure: Number; unit: Dose limiting toxicities
Groups:
- Napabucasin+Sorafenib Phase IB- Dose Level 1: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will be 160 mg twice daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Napabucasin in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Napabucasin+Sorafenib Phase IB- Dose Level 2: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will be 240 mg twice daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Napabucasin in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Amcasertib+Sorafenib Phase IB- Dose Level 1: Amcasetib will be administered orally once daily in combination with sorafenib. The dose of Amcasertib to be administered will be 100mg once daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Amcasertib in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Amcasertib+ Sorafenib Phase IB Dose Level 2: Amcasertib will be administered orally once daily in combination with sorafenib. The dose of Amcasertib will be 200mg once daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Amcasertib in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
Arm/Group | Napabucasin+Sorafenib Phase IB- Dose Level 1 | Napabucasin+Sorafenib Phase IB- Dose Level 2 | Amcasertib+Sorafenib Phase IB- Dose Level 1 | Amcasertib+ Sorafenib Phase IB Dose Level 2
Number analyzed (Participants) | 5 | 10 | 4 | 9
Dose limiting toxicities | 0 | 0 | 0 | 0

2. Primary Outcome: To Assess the Number of Patients Who Experienced Adverse Events for Phase IB.
Description: Assessment of safety of either BBI608 or BBI503 given in combination with sorafenib to patients with hepatocellular carcinoma by reporting of adverse events and serious adverse events
Time Frame: Adverse events will be assessed at baseline, while the participant is taking drugs, and for 30 days after stopping therapy. It was expected that patients would receive between 4-24 weeks treatment.
Measure: Number; unit: count of participants
Groups:
- Napabucasin+Sorafenib Phase IB- Dose Level 1: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will be 160mg twice daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Napabucasin in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Napabucasin+Sorafenib Phase IB - Dose Level 2: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will be 240 mg twice daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Napabucasin in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Amcasertib +Sorafenib Phase IB- Dose Level 1: Amcasetib will be administered orally once daily in combination with sorafenib. The dose of Amcasertib to be administered will be 100mg once daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Amcasertib in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Amcasertib+ Sorafenib Phase IB- Dose Level 2: Amcasetib will be administered orally once daily in combination with sorafenib. The dose of Amcasertib to be administered will be 200mg once daily. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Amcasertib in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
Arm/Group | Napabucasin+Sorafenib Phase IB- Dose Level 1 | Napabucasin+Sorafenib Phase IB - Dose Level 2 | Amcasertib +Sorafenib Phase IB- Dose Level 1 | Amcasertib+ Sorafenib Phase IB- Dose Level 2
Number analyzed (Participants) | 5 | 10 | 4 | 9
count of participants
  Patients with TEAEs | 5 | 10 | 4 | 9
  Patients with TEAEs CTCAE ≥Grade 3 TEAEs | 3 | 8 | 3 | 5
  Patients with serious TEAEs | 0 | 3 | 2 | 5
  Patients with TEAEs leading to treatment discontinuation | 0 | 2 | 2 | 1
  Patients with TEAEs leading to Death | 0 | 0 | 1 | 1
  Patients with TEAEs leading to Napabucasin reduction | 1 | 3 | 0 | 0
  Patients with TEAEs leading to Amcasertib dose reduction | 0 | 0 | 0 | 0
  Patients with TEAEs leading to Napabucasin dose held | 1 | 7 | 0 | 0
  Patients with TEAEs leading to Amcasertib dose held | 0 | 0 | 2 | 6

3. Primary Outcome: Determination of the Recommended Phase II Dose for Napabucasin and Amcasertib Arm in Combination With Sorafenib
Description: To determine the recommended phase II dose for Napabucasin and Amcasertib arm in combination with sorafenib
Time Frame: 16 weeks including 2-week Sorafenib run-in period prior to initiation of combination therapy
Measure: Number; unit: mg
Groups:
- Napabucasin+Sorafenib Phase IB: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will depend on the assigned dose-level cohort. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Napabucasin in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Amcasertib+ Sorafenib Phase IB: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will depend on the assigned dose-level cohort. The patients are considered evaluable for the determination dose level toxicities and determination of dose escalation if they have been exposed to at least 28 days of continues daily administration of Amcasertib in combination with sorafenib at a compliance level of at least 80% Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
Arm/Group | Napabucasin+Sorafenib Phase IB | Amcasertib+ Sorafenib Phase IB
Number analyzed (Participants) | 15 | 13
mg
  Recommended Dose of Napabucasin for phase II | 480 | NA — The recommended dose for Napabucasin and Amcasertib has been evaluated by arm only for phase IB.
  Recommended dose of Amcasertib for Phase II | NA — The recommended dose for Napabucasin and Amcasertib has been evaluated by arm only for phase IB. | 100

4. Primary Outcome: Assessment of Objective Response Rate in the Intent to Treat Population - Phase II
Description: To evaluate the preliminary anti-tumor activity in patients with advanced hepatocellular carcinoma randomized to receive treatment with sorafenib in combination with Napabucasin or sorafenib in combination with Amcasertib, or sorafenib alone; Napabucasin and Amcasertib will be administered at their respective RP2D dose levels for combination administration with sorafenib, which were determined during the phase Ib portion of the study.
  The radiologic assessments will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST for patients with hepatocellular carcinoma.
  ORR was defined as the percentage of patients with a best overall response (BOR) of complete response (CR) or partial response (PR), using both RECIST and mRECIST assessment data.
Time Frame: Assessment of the preliminary anti-tumor activity by performing tumor assessments at baseline and every 8 weeks after the date of the first dose of protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Napabucasin +Sorafenib Phase II | Experimental Amcasertib+Sorafenib Phase II | Sorafenib Phase II
Number analyzed (Participants) | 28 | 10 | 31
percentage of participants
  Assessment of Objective Response Rate based on RECIST 1.1 criteria | 3.6 [0.1 to 18.3] | 0 [0.0 to 30.8] | 9.7 [2.0 to 25.8]
  Assessment of Objective Response Rate based on mRECIST 1.1 criteria | 3.6 [0.1 to 18.3] | 0 [0.0 to 30.8] | 6.5 [0.8 to 21.4]

5. Primary Outcome: Assessment of Disease Control Rate in the Intent to Treat Population- Phase II
Description: To evaluate the preliminary anti-tumor activity in patients with advanced hepatocellular carcinoma randomized to receive treatment with sorafenib in combination with Napabucasin, sorafenib in combination with Amcasertib*, or sorafenib alone; Napabucasin and Amcasertib will be administered at their respective RP2D dose levels for combination administration with sorafenib, which were determined during the phase Ib portion of the study.
  The radiologic assessments will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST for patients with hepatocellular carcinoma.
  Disease control rate (DCR), defined as the proportion of patients with best response of complete response (CR), Partial Response (PR), or stable disease (SD)
Time Frame: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Napabucasin +Sorafenib Phase II | Experimental Amcasertib+Sorafenib Phase II | Sorafenib Phase II
Number analyzed (Participants) | 28 | 10 | 31
percentage of participants
  Assessment of Objective Response Rate based on RECIST 1.1 criteria | 35.7 [18.6 to 55.9] | 70.0 [34.8 to 93.3] | 48.4 [30.2 to 66.9]
  Assessment of Objective Response Rate based on mRECIST 1.1 criteria | 35.7 [18.6 to 55.9] | 50.0 [18.7 to 81.3] | 48.4 [30.2 to 66.9]

6. Secondary Outcome: Assessment of the Pharmacokinetic Profile (Maximum Plasma Concentration and Area Under the Curve) of Either Napabucasin or Amcasertib.
Description: To determine the pharmacokinetic (PK) profile of napabucasin administered in combination with sorafenib and of amcasertib administered in combination with sorafenib.
Time Frame: On Day 15 of the first cycle and Day 15 of the second cycle, prior to dosing and every one hours to 11 hours and 24 hours after first dose
Population: PK parameters were not calculated for this study and are not available. The analyses were not performed as decisions were made to discontinue all clinical development of amcasertib, and of napabucasin for hepatocellular carcinoma.
Groups:
- Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 1: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will be 160mg daily.
  Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug
- Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 2: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin will be 240 mg twice daily Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcsertib Plus Sorafenib Phase IB- Dose Level 1: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 100mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasetib Plus Sorafenib Phase IB- Dose Level 2: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 200mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Napabucasin Plus Sorafenib Phase II: Phase II Napabucasin will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug
- Experimental Amcasertib Plus Sorafenib Phase II: Phase II Amcasertib will be administered in combination with sorafenib at the RP2D determined during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
Arm/Group | Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 1 | Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 2 | Experimental Amcsertib Plus Sorafenib Phase IB- Dose Level 1 | Experimental Amcasetib Plus Sorafenib Phase IB- Dose Level 2 | Experimental Napabucasin Plus Sorafenib Phase II | Experimental Amcasertib Plus Sorafenib Phase II | Sorafenib Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Assessment of the Pharmacodynamic Studies as Well as the Concentration of Study Drug (Either Napabucasin or Amcasertib) in Tumors
Description: To perform biomarker studies for napabucasin administered in combination with sorafenib and for amcasertib administered in combination with sorafenib.
Time Frame: On day 15 of the second cycle
Population: PD assessments were not performed for this study and are not available. Archival tissue, with raw staining scores, and no correlative analyses with clinical data were performed. Analyses were not performed as decisions were made to discontinue all clinical development of amcasertib, and also to discontinue development of napabucasin for hepatocellular carcinoma.
Groups:
- Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 1: Napabucasin will be administered orally twice daily in combination with sorafenib. The dose of Napabucasin to be administered will be 160mg twice daily.
  Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug
- Experimental Amcasertib Plus Sorafenib Phase IB- Dose Level 1: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 100mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
- Experimental Amcasertib Plus Sorafenib Phase IB- Dose Level 2: Amcasertib will be administered orally daily in combination with sorafenib. The dose of Amcasertib to be administered will be 200mg once daily. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose). This dose of sorafenib will be the same for each arm and for each dose-level cohort. Sorafenib should be taken on an empty stomach, one hour prior to or two hours after meals. Sorafenib should not be taken with study drug, and at least 2 hours should separate a dose of sorafenib from a dose of study drug.
Arm/Group | Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 1 | Experimental Napabucasin Plus Sorafenib Phase IB- Dose Level 2 | Experimental Amcasertib Plus Sorafenib Phase IB- Dose Level 1 | Experimental Amcasertib Plus Sorafenib Phase IB- Dose Level 2 | Experimental Napabucasin Plus Sorafenib Phase II | Experimental Amcasertib Plus Sorafenib Phase II | Sorafenib Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of the first treatment until 30 days of the last administration of the study drug for an average period of 28 weeks. The total period for both phase I and phase II of the study was 5 years.
Description: Napabucasin+Sorafenib Phase II:There were 25 who received at least 1 dose.5 discontinued during the Run-inperiod consisting of sorafenib only;total to receive both napabucasin + sorafenib was 20. Amcasertib+Sorafenib Phase II: There were 10 patients and 3 discontinued during the Run-inperiod consisting of sorafenib only;total to receive both amcasertib + sorafenib was 7.Sorafenib Phase II:Patients from napabucasin and amcasertib arms who only received sorafenib were analyzed with sorafenib arm.
Groups:
- Experimental Napabucasin+Sorafenib Phase IB- Dose Level 1; Experimental Napabucasin +Sorafenib Phase IB- Dose Level 2: Patients who have received at least one dose of Napabucasin in combination with sorafenib during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Experimental Amcasertib+Sorafenib Phase IB- Dose Level 1; Experimental Amcasertib+Sorafenib Phase IB- Dose Level 2: Patients who have received at least one dose of Amcasertib in combination with sorafenib during the phase 1 dose-escalation portion of study. Sorafenib will be administered at a fixed dose of 400 mg twice daily (800 mg total daily dose).
- Experimental Napabucasin +Sorafenib Phase II: Phase II: Patients who have received at least one dose of Napabucasin (at the RP2D determined for napabucasin plus sorafenib during the Phase 1b portion) in combination with sorafenib. In the amcasertib + sorafenib arm, there were 10 patients randomized. Of these 10 patients, 3 discontinued during the Run-in period consisting of sorafenib monotherapy; therefore, the total to receive both amcasertib + sorafenib in Phase 2 was 7
- Experimental Amcasertib +Sorafenib Phase II: Phase II: Patients who have received at least one dose of amcasertib (at the RP2D determined for amcasertib plus sorafenib during the Phase 1b portion) in combindation with sorafenib. There were 28 total randomized and 25 who received at least 1 dose of study treatment. Of these 25 patients, 5 discontinued during the Run-in period consisting of sorafenib monotherapy; therefore, the total number of patients to receive both napabucasin + sorafenib in Phase 2 was 20
- Sorafenib Phase II: Phase II: Patients who have received at least one dose of sorafenib
Arm/Group | Experimental Napabucasin+Sorafenib Phase IB- Dose Level 1 | Experimental Napabucasin +Sorafenib Phase IB- Dose Level 2 | Experimental Amcasertib+Sorafenib Phase IB- Dose Level 1 | Experimental Amcasertib+Sorafenib Phase IB- Dose Level 2 | Experimental Napabucasin +Sorafenib Phase II | Experimental Amcasertib +Sorafenib Phase II | Sorafenib Phase II
All-Cause Mortality (participants affected / at risk) | 4/5 | 7/10 | 4/4 | 9/9 | 15/20 | 6/7 | 23/36
Serious Adverse Events (participants affected / at risk) | 0/5 | 3/10 | 2/4 | 5/9 | 10/20 | 3/7 | 16/36
Other Adverse Events (participants affected / at risk) | 5/5 | 10/10 | 4/4 | 9/9 | 20/20 | 7/7 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Napabucasin+Sorafenib Phase IB- Dose Level 1 (N=5) | Experimental Napabucasin +Sorafenib Phase IB- Dose Level 2 (N=10) | Experimental Amcasertib+Sorafenib Phase IB- Dose Level 1 (N=4) | Experimental Amcasertib+Sorafenib Phase IB- Dose Level 2 (N=9) | Experimental Napabucasin +Sorafenib Phase II (N=20) | Experimental Amcasertib +Sorafenib Phase II (N=7) | Sorafenib Phase II (N=36)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 2 | 3
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Esophageal varices (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute Focal Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gastointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small bowel obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary Track infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Altered mental status (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia generalized (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoxia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary tube displaced (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile Sten Occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mature B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Napabucasin+Sorafenib Phase IB- Dose Level 1 (N=5) | Experimental Napabucasin +Sorafenib Phase IB- Dose Level 2 (N=10) | Experimental Amcasertib+Sorafenib Phase IB- Dose Level 1 (N=4) | Experimental Amcasertib+Sorafenib Phase IB- Dose Level 2 (N=9) | Experimental Napabucasin +Sorafenib Phase II (N=20) | Experimental Amcasertib +Sorafenib Phase II (N=7) | Sorafenib Phase II (N=36)
Diarrhea (Gastrointestinal disorders) | 4 | 7 | 3 | 7 | 17 | 6 | 18
Nausea (Gastrointestinal disorders) | 3 | 5 | 2 | 5 | 9 | 3 | 17
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 3 | 10 | 3 | 7
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 5 | 4 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 4 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 8
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 8 | 1 | 6 | 15 | 6 | 22
Asthenia (General disorders) | 0 | 5 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrosaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 2 | 3 | 3 | 9
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 2 | 5 | 8 | 3 | 16
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotrasnferase increased (Investigations) | 1 | 3 | 0 | 0 | 5 | 2 | 6
Weight Decreased (Investigations) | 2 | 2 | 1 | 3 | 4 | 3 | 14
Blood bilirubin increased (Investigations) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 1 | 2 | 5 | 1 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of any proposed publication or disclosure of the results of the Study will be given to Sponsor for review at least thirty (30) days prior to the date of submission for publication ( including abstracts) or of public disclosure ( the review period).

DOCUMENTS (2):
  • Study Protocol (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02279719/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT02279719/SAP_001.pdf